CLINICAL TRIAL: NCT01763528
Title: High Protein Diet , CRP and CVD Risk Factors
Brief Title: High Protein Weight Loss Diet, High Sensitivity C-Reactive Protein and Cardiovascular Risks Among Obese Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences,, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: high protein in women
Record Dates: First submitted 2012-12-18; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Body Mass Index Quantitative Trait Locus 8 Disorder; Tangier Disease
Keywords: body weight; Low-density-lipoprotein-type
MeSH Terms: conditions — Tangier Disease; Body Weight | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nutrition intervention (Active Comparator): high protein diet
  Interventions: Other: nutrition intervention
- control group (No Intervention): control diet

INTERVENTIONS:
Other: nutrition intervention — high protein diet
  Arms: nutrition intervention

SUMMARY:
The investigators aimed to determine the effects of HP diet on CVD risk factors and hs-CRP among overweight and obese women.

DETAILED DESCRIPTION:
Background: Studies regarding the effects of high protein (HP) diet on cardiovascular (CVD) risk factors have reported contradictory results.

Objective: In present study, we aimed to determine the effects of HP diet on CVD risk factors and hs-CRP among overweight and obese women.

Design: In this randomized controlled trial, we recruited 60 overweight and obese women, aged 20-65 years into HP or control energy restricted diets for three months (protein, carbohydrate, fat: 25%, 45%, 30% vs. 15%, 55%, 30%, respectively). Total protein amount, divided to animal and plant sources in 50%-50% and animal sources distributed (half/half) between meats and dairy products. Fasting blood samples, hs-CRP, lipid profile, systolic and diastolic blood pressure and anthropometric measurements were measured based on the standard guidelines.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 20-65 years
* BMI > 25 kg/m2
* were no smoker
* no history of renal, liver, metabolic diseases or type 1 or 2 diabetes

Exclusion Criteria:

* had gastrointestinal, respiratory, cardiovascular, metabolic, liver and renal -diseases
* had macroalbuminuria
* were pregnancy or lactating

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
the amount of weight reduction in two dietary groups | 3 months
  weight reduction (kg)

SECONDARY OUTCOMES:
LDL-C (mg/dl | 3 months
  measurement of LDL-C (mg/dl), HDL-C (mg/dl), total cholesterol (mg/dl), fasting blood glucose (mg/dl), systolic and diastolic blood pressure (mmHg), c reactive protein by the measurement of blood samples.
HDL-C (mg/dl) | 3 months
total cholesterol (mg/dl) | 3 months
fasting blood glucose(mg/dl) | 3 months
blood pressure (mmHg) | 3 months
C-reactive protein (mc/dl) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfan University of Medical Sciences

REFERENCES:
- [Derived] Azadbakht L, Izadi V, Surkan PJ, Esmaillzadeh A. Effect of a High Protein Weight Loss Diet on Weight, High-Sensitivity C-Reactive Protein, and Cardiovascular Risk among Overweight and Obese Women: A Parallel Clinical Trial. Int J Endocrinol. 2013;2013:971724. doi: 10.1155/2013/971724. Epub 2013 Aug 6. PMID 23986778